CLINICAL TRIAL: NCT05639179
Title: An Investigator-initiated Trial to Evaluate the Efficacy and Safety of Anti-CD19 Universal CAR-T Cells in the Treatment of Relapsed/Refractory(r/r) CD19+ B-cell Acute Lymphoblastic Leukemia(B-ALL)
Brief Title: Novel Anti-CD19 Universal CAR-T Cells for r/r CD19+ B-ALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM-010
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-ALL
Keywords: universal CAR-T(UCAR-T); CD19
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of UCAR-T Cells after lymphodepletion.
  Interventions: Biological: UCAR-T Cells

INTERVENTIONS:
Biological: UCAR-T Cells — UCAR-T Cellswill be administered by vein. The trial includes two portions. The first portion is a"3+3"dose escalation study, in which three dose groups are set:Dose level one:1×10^6 cells/kg;Dose level two:2×10^6 cells/kg;Dose level three:5×10^6 cells/kg. Each dose group requires at least three subjects. The trial will start from dose level one. The second portion includes a dosage extended cohort and will start after the finish of the"3+3"dose escalation study. Twelve subjects will get infusion of UCAR-T Cells at the best dose verified in the first portion.

SUMMARY:
This is a single-arm, single-center, open-labeled clinical study to evaluate the safety and efficacy of UCAR-T Cells injection for patients with relapsed/refractory(r/r) B-cell Acute Lymphoblastic Leukemia(B-ALL).

DETAILED DESCRIPTION:
Although the anti-CD19 CAR-T cell therapies have gained significant clinical outcome in patients with r/r B-ALL，autologous CAR-T is not feasible for some patients. To make further improvement, the investigators are going to conduct a clinical trial using universal CAR-T(UCAR-T) cells targeting CD19 for r/r B-ALL patients.

After enrollment, patients will get a 3-5 days lymphodepletion therapy, then the UCAR-T Cells will be infused by vein. Subjects will be followed for safety and efficacy up to 12 weeks. For those with a durable remission 12 weeks after infusion, the follow-up will last for at least 12 months for disease control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 2-75 years;
2. A definite diagnosis of relapsed/refractory B-ALL and a percentage of primitive/naive lymphocytes >5% in bone marrow at baseline (flow cytometry);
3. CD19 expression was positive in bone marrow or peripheral blood tumor cells;
4. ECOG score 0-2 points;
5. Expected survival time ≥3 months;
6. Adequate liver, kidney, heart and lung function;
7. Patients who have recovered from acute toxic effects of prior chemotherapy should be excluded from the trial at least one week apart;
8. Women of childbearing age have negative blood pregnancy test before the start of the trial, and agree to take effective contraceptive measures during the trial until the last follow-up; male subjects with partners of childbearing potential agree to take effective contraceptive measures during the trial until the last follow-up;
9. Voluntarily sign the informed consent.

Exclusion Criteria:

1. Presence of other concurrent active malignancy;
2. People with severe mental disorders;
3. A history of any of the following genetic disorders, such as Fanconi anemia, Schu-Day syndrome, Gerstmann syndrome, or any other known bone marrow failure syndrome;
4. Acute GVHD of grade II-IV or extensive chronic GVHD;
5. Had grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other clinically prominent heart disease within one year prior to enrollment;
6. The presence of any indwelling catheter or drainage (e.g., percutaneous nephrostomy, indwelling catheter, bile drainage, or pleural/peritoneal/pericardial catheter), except for patients who are permitted to use dedicated central venous catheters;
7. A history or disease of the central nervous system(CNS), such as seizure disease, cerebrovascular ischemia/bleeding, dementia, cerebellar disease, or any autoimmune disease involving the CNS;
8. Human immunodeficiency virus (HIV) seropositivity; Hepatitis B surface antigen positive or hepatitis B core antibody positive, and HBV-DNA positive; Patients with hepatitis C (HCV-RNA quantitative test results positive); Or the presence of other serious active viral or bacterial infections or uncontrolled systemic fungal infections;
9. Patients with severe history of allergy or allergic constitution;
10. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) leading to end-organ damage or requiring systemic immunosuppressive/systemic disease modulating drugs within the past 2 years;
11. Had or is suffering from interstitial lung disease (e.g., pneumonia, pulmonary fibrosis);
12. Had undergone other clinical trials in the 4 weeks prior to participating in this trial;
13. Poor compliance due to physiological, family, social, geographical and other factors, unable to cooperate with the study protocol and follow-up plan;
14. For patients contraindicated with cyclophosphamide and fludarabine chemotherapy;
15. Subjects requiring systemic corticosteroid therapy (prednisone ≥5mg/ day or equivalent dose of another corticosteroid) or other immunosuppressive agents within 1 month after UCAR-T cell reinfusion, except for adverse events;
16. Receiving donor lymphocyte infusion within 6 weeks before enrollment;
17. Pregnant and lactating women;
18. Any other condition that the investigator deemed inappropriate for inclusion.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after infusion
  Neurotoxicity and/or CRS≥G3.
Incidence of Treatment Related adverse events (AEs) | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
Persistence of CAR-T cells | Up to 24 weeks after infusion
  The persistence over time of CAR-T cells in the peripheral blood as determined by flow cytometry and qPCR.
Objective response rate (ORR) | At 4,8,12 weeks after infusion
  Patients who achieve CR(complete response) or CRi after infusion
Progression-free survival (PFS) | Up to 24 weeks after infusion
  Progression-free survival (PFS) is the time between the time a patient with tumor disease receives treatment and the time between the observation of disease progression or death from any cause.
Overall survival (OS) | Up to 24 weeks after infusion
  Overall survival (OS) is the time from randomization to death from any cause.
Duration of remission (DOR) | Up to 24 weeks after infusion
  Duration of remission (DOR) is the time from the first detection of CR or PR to the discovery of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Sanbin, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China